CLINICAL TRIAL: NCT00682097
Title: A Randomized, Double-Blind, Multiple-Ascending-Dose, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO4998452 Following Oral Administrations in Patients With Type 2 Diabetes Mellitus
Brief Title: A Multiple Ascending Dose Study of RO4998452 in Patients With Type 2 Diabetes Mellitus.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BP21549; 2007-007120-18
Record Dates: First submitted 2008-05-20; First posted 2008-05-22 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (7):
- 1 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 2 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 3 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 4 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 5 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 6 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo
- 7 (Experimental)
  Interventions: Drug: RO4998452; Drug: placebo

INTERVENTIONS:
Drug: RO4998452 — Escalating oral doses
Drug: placebo — Oral doses

SUMMARY:
This study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of multiple ascending doses of RO4998452 compared to placebo in patients with type 2 diabetes mellitus. Successive cohorts of patients will be randomized to receive either active drug, at escalating doses, or placebo. The anticipated time on study treatment is <3 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18-65 years of age;
* type 2 diabetes;
* either treated by diet and exercise alone or with metformin.

Exclusion Criteria:

* type 1 diabetes mellitus;
* uncontrolled hypertension;
* clinically severe diabetic complications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2008-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
AEs, laboratory parameters, vital signs. | Throughout study
AUC0-24h, Cmax | Days 1 and 14

SECONDARY OUTCOMES:
Parameters of glucose metabolism | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (3):
- United States (2):
  - Chula Vista, California
  - San Antonio, Texas
- Neuss, Germany